CLINICAL TRIAL: NCT01189565
Title: Continuous Postoperative Pulse Oximetry in Patients Presenting for Total Hip and Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Matthew D. McEvoy, MUSC
Other Study IDs: HR-19772
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2010-08

CONDITIONS: Total Knee Replacement
Keywords: Total Hip Replacement/Revision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Joint Replacement Patients

SUMMARY:
The purpose of this study is to evaluate the incidence of low levels of oxygen as determined by standard pulse oximetry monitor in patients who have had total hip or knee replacement/revision.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing knee replacement or hip replacement/revision

Exclusion Criteria:

* Patients requiring mechanical ventilation after surgery
* Patients with hemoglobinopathy that cause inaccurate pulse oximetry

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Joint Replacement
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D McEvoy, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC, Charleston, South Carolina, United States

REFERENCES:
- [Background] Lawrence VA, Cornell JE, Smetana GW; American College of Physicians. Strategies to reduce postoperative pulmonary complications after noncardiothoracic surgery: systematic review for the American College of Physicians. Ann Intern Med. 2006 Apr 18;144(8):596-608. doi: 10.7326/0003-4819-144-8-200604180-00011. PMID 16618957
- [Background] McAlister FA, Bertsch K, Man J, Bradley J, Jacka M. Incidence of and risk factors for pulmonary complications after nonthoracic surgery. Am J Respir Crit Care Med. 2005 Mar 1;171(5):514-7. doi: 10.1164/rccm.200408-1069OC. Epub 2004 Nov 24. PMID 15563632
- [Background] Lawrence VA, Hilsenbeck SG, Mulrow CD, Dhanda R, Sapp J, Page CP. Incidence and hospital stay for cardiac and pulmonary complications after abdominal surgery. J Gen Intern Med. 1995 Dec;10(12):671-8. doi: 10.1007/BF02602761. PMID 8770719